CLINICAL TRIAL: NCT01481090
Title: Electro-acupuncture and Assisted Reproductive Technology: Impact of EA on Endometrium During Medicated Frozen Embryo Transfer Uterine Preparation
Brief Title: Electro-acupuncture and Assisted Reproductive Technology
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB violations
Sponsor: National University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NUHS H1007
Record Dates: First submitted 2011-11-22; First posted 2011-11-29 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Infertility
Keywords: Infertility; acupuncture; frozen embryos; endometrium; TCM
MeSH Terms: conditions — Infertility | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electro-Acupuncture (Active Comparator): Group will receive 4 acupuncture treatments over 14 days during hormone treatment
  Interventions: Procedure: Acupuncture, Electro-Acupuncture
- Control (No Intervention): Group will not receive acupuncture.

INTERVENTIONS:
Procedure: Acupuncture, Electro-Acupuncture — Participants will receive 4 Electro-acupuncture stimulation applied to acupoints SP-6, Zi-Gong, CV-3 and CV-4acupuncture treatments during hormone treatment.
  Arms: Electro-Acupuncture

SUMMARY:
One of the most widely used procedures in reproductive medicine technologies is In Vitro Fertilization (IVF). During the IVF procedure, there are sometimes unused embryos that are frozen to be used at later times. If these embryos are thawed and transferred back to the mother, proper development of the uterine lining plays an important role in outcome of pregnancy. Electro-acupuncture (EA), a technique where electrical current is applied to the needle to stimulate an acupoint, has been shown to increase uterine blood flow, increasing the likelihood of developing a more ideal endometrial lining. This randomized study aims to evaluate the impact of EA on endometrium undergoing medicated frozen embryo transfer cycle preparation. The treatment group will receive four acupuncture treatments during the medicated uterine preparation. Endometrial thickness will be compared to a group that does not receive acupuncture.

DETAILED DESCRIPTION:
All the subjects in the study will be randomized and their participation is completely voluntary. Patients recruited to join the study will not receive any monetary compensation for participation.

This research will include 100 female subjects, ages 21-45, undergoing medicated frozen embryo transfer (mFET). The subjects will be randomized into treatment and the non-treatment groups. The non-treatment group will undergo the medicated uterine preparation for FET according to the fertility clinic's protocol.

Subjects in the treatment group will receive four electro-acupuncture (EA) treatments in addition to the mFET protocol, starting after the 1st Ultrasound measurement which constitutes as a baseline, until the start of the progesterone administration. Endometrial thickness will be measured using ultrasound and estrogen (E2) levels will be measured by blood samples as a standard measure to assess the time of P4 (progesterone) supplementation. This step will be done by the participant's fertility clinic according to the clinic's protocol.

Acupuncture points of LI-4, LV-3, SP-6, Zi Gong, CV-3, CV-4, ST-36 will be needled. Electro-stimulation will be applied to acupoints SP-6, Zi-Gong, CV-3 and CV-4 at low frequency. The needle retention with electro-stimulation will last for 25 minutes. After the 25 minutes, the needles and the electro-stimulation will be removed and the patients will be dismissed.

Ultrasound results measuring endometrium will be obtained from the subject's fertility clinic. US and bloodwork will be performed at baseline, and before the progesterone administration according to the fertility clinic. This US measurement and bloodwork results will be used for statistical analysis to compare endometrial lining of the two groups. The final discussion will be presented according to the findings.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing medicated frozen embryo transfer uterine preparation
* Ages between 21-45 years old
* Must be fluent in English
* Must be willing to receive four electro-acupuncture treatments
* Must be willing to provide access to medical records from the fertility clinic

Exclusion Criteria:

* Males
* Subjects involved with fresh IVF cycle
* Subjects with pace maker
* Subjects with history of seizure disorders
* All others who do not meet the inclusion criteria

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Change in endometrium thickness during hormone treatment | Baseline, day 8 and day 15 of hormone treatment
  As part of the preparation for embryo transfer, patients undergo ultrasound during hormone treatment to assess endometrium thickness. Research participants will agree to release ultrasound results to the research personnel to determine whether acupuncture treatments affect endometrium thickness compared to no acupuncture treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Y Cai, Ph.D, Principal Investigator — National University of Health Sciences
Locations (2):
- United States (2):
  - Tiffani Kim Institute, Chicago, Illinois
  - National University of Health Sciences, Lombard, Illinois